CLINICAL TRIAL: NCT00211250
Title: An Exploratory Study Comparing Compliance, Tolerability, Efficacy and Adverse Events in Bipolar I and II Patients From Valproic Acid to Depakote ER
Brief Title: Comparing Compliance, Tolerability, Efficacy and Adverse Events in Bipolar Tients From Valproic Acid to Depakote ER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Joliet Center for Clinical Research (Other)
Collaborators: Abbott (Industry)
Responsible Party: Cosme o. lozano, MD, Joliet Center for Clinical research
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JCCR-001
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2009-01-28 (Estimated); Status verified 2009-01

CONDITIONS: Mood Disorder
Keywords: Depakote Er and Valproic Acid
MeSH Terms: conditions — Mood Disorders | interventions — Valproic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Valproic Acid and Depakote ER

SUMMARY:
The purpose of this study is to compare compliance, tolerability, effectiveness, and side-effects in Bipolar I and II patients switching from Valproic Acid to Depakote ER.

DETAILED DESCRIPTION:
Over the next year between 20 and 40 patients, who meet all inclusion and exclusion criteria, will be entered into the study. The treatment period of the study will last at least 10-13 weeks depending on how quickly your Depakote ER level reaches a therapeutic level (50-100mcg/mL).

At your first visit:

* A medical and psychiatric history will be obtained. For your own safety, it is your responsibility to tell the study doctor or study staff of your past and present diseases, all allergies and medical conditions, and all medications that you currently or recently have taken, including over-the-counter medications such as vitamins, allergy medicines, and herbal drugs. A physical examination and vital signs, which will include measuring your height, weight, blood pressure, respiratory (breathing) rate, and heart rate (pulse).
* Blood samples will be taken, through a needle in your vein. Approximately 2-2 ½ tablespoons (28 or 38 ml) of blood for routine testing of hematology (red and white blood cells) and clinical chemistry (blood salt, sugar, fats, and hormones, and tests of liver, kidney and thyroid function), and valproate level
* A urinalysis, a urine pregnancy test (for all females), and a urine drug screen will be obtained. If you are a woman and your urine pregnancy test is positive, a blood test will be done to confirm this; you will not be able to participate in this study if this is also positive.
* An electrocardiogram (ECG - a painless electrical tracing of your heart function).
* Psychiatric scales designed to measure past compliance, side-effects, and your bipolar symptoms will be administered. (See the Attached Schedule of Events for a list of all Procedures required during the study) Patients, who continue to meet all inclusion and exclusion criteria, will return for a baseline visit (Visit 2). At this visit you will discontinue valproic acid and begin taking Depakote ER the following day. The total daily dose will be adjusted to be 8-20% higher than your original valproic acid dose, at the discretion of the Investigator, in order to reach therapeutic levels. Rating scales will be administered and the study drug (Depakote ER) will be dispensed.

Your study doctor or staff will explain the amount of medication you will receive, and will give you instructions on how to take it. It is important that your study drug is not taken by anyone else. Your study doctor and other study staff, whom you are to ask any questions about the study drug's effects and any side effects, will regularly check your response to treatment. If you get worse, the study drug dose may be changed, or you may be given additional medications, or the study drug may be stopped and you will be given another drug instead.

Before continuing to visit 3 you must reach a valproate level of 50-100mcg/mL. Weekly titration visits (T1-T4) will be scheduled and blood samples will be taken to test the Valproic level in your blood. The study doctor may adjust your dose, until a level of 50-100 mcg/ml is reached. If the above level is not reached within four weeks of visit 2, you will be discontinued from the study.

After the therapeutic level is reached, you will be asked to return in one week for visit 3, four weeks for visit 4, and another four weeks for the final visit, visit 5. Overall, your treatment with Depakote ER will be between 10-13 weeks in duration. During visits 3 and 4 the Depakote ER dose may be adjusted in 250mg or 500mg increments to maintain adequate level, to manage side effects and/or manage bipolar symptoms at the discretion of the study doctor. In addition, you will be asked to report any side effects and complete the psychiatric scales at each visit and blood samples will be taken at visits 3 and 5. (See the Schedule of Events for more details)

ELIGIBILITY:
Inclusion Criteria:

* Bipolar I and II patients, age 18 and older, currently tolerating a stable dose of Valproic Acid for at least 3 months with a current Valproic Acid level of at least 50 mcg/mL at screening and baseline,

Exclusion Criteria:

* Women who are pregnant or breast feeding or intending to become pregnant, contraindication or history of hypersensitivity to valproic acid, DVPX or DVPX ER.
* Clinically significant organ disease, clinically significant abnormalities in physical examination, EKG, or lab test, history of any disease which in the investigator's opinion may confound the results of the study or pose additional risk.
* Other principle nonpsychotic or psychotic psychiatric diagnosis. Patients weighing >300 pounds.
* Patients taking any other mood stabilizers.
* Patients not already on a stable dose of valproic acid or have a Valproic Acid level less than 50 mcg/mL at screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2005-07; Primary Completion 2006-07 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Primary Measure: Safety and Tolerability.
Comparisons will be made between baseline and final measures of adverse events and UKU results.

SECONDARY OUTCOMES:
Secondary Measures: Compliance and efficacy.
Comparison of YMRS and MADRS scores

CONTACTS AND LOCATIONS:
Overall Officials: Cosme O Lozano, M.D., Principal Investigator — JCCR
Locations (1):
- Cosme Lozano M.D., Joliet, Illinois, United States

REFERENCES:
- [Background] Berk, M & Berk, L. (2004). Mood stabilizers and treatment adherence in bipolar disorder: addressing adverse events. Bowden C.L., Calabrese J.R., McElroy S.L., Gyulai L., Wassef A., Petty F., Pope H.G. Jr, Chou J.C., Keck P.E. Jr, Rhodes L.J., Swann A.C., Hirschfeld R.M., Wozniak P.J., (2000). Valproate in the treatment of acute mania: placebo-controlled study. Archives of General Psychiatry, 48, 62-68. Pope, S. J. (2002). Nonadherence with mood stabilizers: prevalence and predictors. Journal of Clinical Psychiatry, 63, 384-90. Sajatovic, M., Davies M., & Hrouda, D.R. (2004). Enhancement of treatment adherence with patients with bipolar disorder. Psychiatric Services, 55(3), 264-69. Depakote ER package insert, Abbott Laboratories, 2002.
- See also: Research Site — http://www.jccr.net